CLINICAL TRIAL: NCT04771936
Title: Relationship of Core Stability on Pain and Functional Levels in Patients Diagnosed With Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Ilona Dalmas, Principal investigator, University of Malta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2395
Record Dates: First submitted 2021-02-20; First posted 2021-02-25 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Osteoarthritis, Hip
Keywords: Hip; Osteoarthritis; Exercise; Core Stability
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients with a diagnosis of OA hip who are awaiting a total hip replacement will be recruited in this study. Both male and female subjects age 40 years and over will be included in the study.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to the three groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group who shall be awaiting surgery and not receiving a regular physiotherapy exercise intervention
- Conventional Exercise Group (Active Comparator): The conventional exercise group shall be subject to a set of conventional exercises based on a program described by Deyle et al (2000).
  Interventions: Other: Physiotherapy Exercises
- Conventional Exercise Group with added core exercises (Experimental): This exercise group shall be subject to a set of conventional exercises based on a program described by Deyle et al (2000) and core exercises aimed at the activation of the core muscles as adapted from Imai et al (2010).
  Interventions: Other: Physiotherapy Exercises

INTERVENTIONS:
Other: Physiotherapy Exercises — All patients shall be randomly assigned to 3 groups: the control group who shall be awaiting surgery and not receiving a regular physiotherapy, the exercise group who shall be subject to a set of conventional exercises and a core exercise group who shall be performing the conventional exercises plus exercises aimed at the activation of core muscles. These exercises shall be carried out 3 times weekly for a period of 3 months. During the first 4 weeks, all sessions shall be supervised by a physiotherapist. From the 5th to the 8th week, patients shall attend 2 supervised sessions and complete the 3rd one at home. Between the 9th and the 12th week, patients shall then attend 1 supervised intervention and complete 2 sessions at home.Patients assigned to the control group shall be given a chance to enrol into the program upon completion of the study if they wish to do so.
  Arms: Conventional Exercise Group; Conventional Exercise Group with added core exercises

SUMMARY:
Osteoarthritis (OA) is a common disease that occurs more commonly amongst the elderly and is caused by the destruction of the joint cartilage. It is considered to be one of the most common joint disorders worldwide and a main cause of disability amongst older adults. After the knee, the hip is considered to be the second most commonly affected joint by OA. One of the functional capacities affected by OA is muscle strength with studies looking into knee OA documenting a decrement of this measure. It is reported that the muscle strength of the quadriceps, hamstrings and other musculature around the hip is significantly impaired in patients with knee OA compared to age-matched controls.

Evidence for quadriceps muscle weakness in knee OA is consistent and programs based on quadriceps strengthening exercises as a core component in the management of knee OA are now evidence-based. Lower extremity muscle weakness is also apparent in hip OA. However, compared to the knee, there is less literature on muscle strength in hip OA with guidelines for therapeutic exercise prescription being more expert rather than evidence-based. Therefore, one of the major questions that arises here is whether muscle weakness as observed in knee OA is evident in hip OA, and if so, which muscles are most affected.

A concept which has been found to help diminish the effect of decreased muscle strength in the above mentioned muscle groups is optimal core stability. Core stability contributes to strength, endurance, flexibility and motor control all of which optimise the stability of the spine during both dynamic and static tasks in daily normal biomechanical function in patients with a diagnosis of OA knees. Despite such evidence, no studies to the knowledge of the researcher have looked into the effects of core stability on pain and functional levels in patients with a diagnosis of OA hip. A lack of literature in relation to this aspect is due to the unavailability of a gold standard for measuring core stability.

Therefore, the objective of this study will be multifold with an investigation into which muscles in the lower limb are predominantly weaker, whether there is core muscle weakness in patients with hip OA, looking for any correlation between both these factors and whether an exercise programme leads to changes on functional activity and pain levels.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common disease that occurs more commonly amongst the elderly and is caused by the destruction of the joint cartilage. It is considered to be one of the most common joint disorders worldwide and a main cause of disability amongst older adults. After the knee, the hip is considered to be the second most commonly affected joint by OA.

One of the functional capacities affected by OA is muscle strength with studies looking into knee OA documenting a decrement of this measure. The muscle strength of the quadriceps, hamstrings and other musculature around the hip is significantly impaired in patients with knee OA compared to age-matched controls.

Evidence for quadriceps muscle weakness in knee OA is consistent and programs based on quadriceps strengthening exercises as a core component in the management of knee OA are now evidence-based. Lower extremity muscle weakness is also apparent in hip OA. However, compared to the knee, there is less literature on muscle strength in hip OA with guidelines for therapeutic exercise prescription being more expert rather than evidence-based. Therefore, one of the major questions that arises here is whether muscle weakness as observed in knee OA is evident in hip OA, and if so, which muscles are most affected.

A concept which has been found to help diminish the effect of decreased muscle strength in the above mentioned muscle groups is optimal core stability. Core stability contributes to strength, endurance, flexibility and motor control all of which optimise the stability of the spine during both dynamic and static tasks in daily normal biomechanical function in patients with a diagnosis of OA knees. Despite such evidence, no studies to the knowledge of the researcher have looked into the effects of core stability on pain and functional levels in patients with a diagnosis of OA hip. Lack of literature in relation to this aspect is due to the unavailability of a gold standard for measuring core stability.

Therefore, the objective of this study will be multifold with an investigation into which muscles in the lower limb are predominantly weaker, whether there is core muscle weakness in patients with hip OA, looking for any correlation between both these factors and whether an exercise programme leads to changes on functional activity and pain levels.

All the patients who give consent to participate shall be randomly assigned to three groups being the control group who shall be awaiting surgery and not receiving a regular physiotherapy exercise intervention, the exercise group who shall be subject to a set of conventional exercises based and a core exercise group who shall be performing the conventional exercises plus exercises aimed at the activation of the core muscles. These exercises shall be carried out three times weekly for a period of three months. During the first four weeks, all sessions shall be supervised by a physiotherapist who shall monitor and increase the duration or difficulty of exercises according to patients' progression. From the 5th to the 8th week, patients shall attend two supervised sessions and complete the third one at home. Between the 9th and the 12th week, patients shall then attend one supervised intervention and complete two exercise sessions at home. All patients shall be given a copy of the exercise sheet with instructions for use at home. Anonymisation shall be ensured with every patient through assignment of a random code for every individual. Patients assigned to the control group shall be given a chance to enrol into the program upon completion of the study if they wish to do so.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting a total hip replacement
* Anyone above the age of 40 years

Exclusion Criteria:

* Patients with neurologic conditions affecting mobility
* Patients with cognitive impairments
* Patients not willing to comply

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain levels assessed using the Numerical Pain Rating Scale (NPRS) | Week 0 and week 12
  The NPRS is a type of pain scale widely used in the clinical setting aswell as in research. The research found that the NPRS is a simple and valid tool to use with Cleland et al (2008) reporting acceptable construct validity for this tool (p < 0.001). It is usually presented on a horizontal line on which the patient's pain intensity is represented by a point between the marks of 0 (no pain) to 10 (extreme pain). The NPRS is a segmented, numerical version of the Visual Analogue Scale (VAS), as shown in the image below. Its simplicity, reliability, and validity make the NPRS the optimal tool for describing pain severity or intensity (The British Pain Society, 2019).
Change in functional Levels assessed using the WOMAC Scale | Week 0 and week 12
  The Western Ontario and McMaster Universities (WOMAC) is a widely used instrument which is specific to assessing patients with hip and knee OA. This assessment tool is self- administered and is multidimensional (Bellamy, 2008). It consists of 33 items which evaluate the health and function of the patient from various aspects including clinical symptoms (5 questions), severity of joint stiffness (2 questions), degree of pain (9 questions), and activity of daily living (17 questions). Each question has five subscales were the subject score between situations of never or none to situations of extreme or always. A higher score is a representation of a better situation and less pain. Different validation studies of WOMAC make this clinical instrument usable for knee and hip OA and enable clinical investigators to assess those clinical outcome reports using this index from different parts of the world collectively (Ebrahimzadeh et al, 2014).
Change in functional Levels assessed using the 6 MWT | Week 0 and week 12
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. Such a test has been reported to be a valid and reliable indicator of aerobic fitness (ATS guidelines, 2002). It is considered to be a useful objective baseline measure and has normative results and minimal clinically important differences established for a range of older individuals. The subjects will be instructed that they may stop and rest during the test, but the time will keep running. At the end of the six minutes, the time walked and distance will be noted and recorded. Standardised encouragement is provided at 1-minute intervals, and the person should not be paced. Individuals may use assistive devices during the test (ATS guidelines, 2002).
Change in lower limb muscle strength | Week 0 and week 12
  All subjects will undergo peak isometric lower limb muscle torque testing for the following muscle groups: Quadriceps, Hamstrings, Adductors and Abductors using a dynamometer. A demonstration on how to carry out the test correctly will be done together with a single trial to familiarise with the participants with the technique and procedure. A maximum of three attempts will be performed with the average result taken. Participants will be instructed to exert maximal effort and will be verbally coached to push as hard as they can for each recorded trial.
Change in core Muscle Strength using a pressure biofeedback unit (PBU) | Week 0 and week 12
  Participants will be placed in a supine position with the pelvis over the pressure biofeedback unit (PBU) and their hands resting over their chest. The PBU will be placed under the lumbar spine at the level of L3, with a pressure of 40 mm Hg. The participants will be asked to place their hip in flexion or their knee in flexion/extension while in the supine position. They will be asked to 'Take a deep breath in and draw their navel in toward their spine as they exhale'. Each participant will be asked to hold the contraction for as long as they can while maintaining the contraction at 40mmHg on the PBU gauge. Those able to maintain the abdominal contraction for at least 10 seconds at 40 mmHg will be considered as having good core strength. Those unable to hold the contraction for 10 seconds at the mentioned pressure will be considered as having a weak core (Rajan Bhore et al, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Tonio Agius, PhD, Study Director — Lecturer at University of Malta
Locations (1):
- Faculty of Health Sciences, Msida, Malta

IPD SHARING:
Plan to Share IPD: No